CLINICAL TRIAL: NCT00656526
Title: Intraoperative Perineural Injection of Lidocaine for Postlaminectomy Pain
Brief Title: Preemptive Analgesia for Postlaminectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Assistant Professor Cengiz Mordeniz, Harran University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 012
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Laminectomy
Keywords: analgesia, postlaminectomy , lidocaine, dorsal root
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A01L (Placebo Comparator)
  Interventions: Drug: Lidocaine, perineural injection, intraoperatively; Drug: Lidocaine
- B01C (No Intervention)

INTERVENTIONS:
Drug: Lidocaine, perineural injection, intraoperatively — 0.5 cc lidocaine, one single injection over the dorsal root.
  Other Names: lidocaine
  Arms: A01L
Drug: Lidocaine — 0.5 cc %2 lidocaine,single injection
  Arms: A01L

SUMMARY:
To relieve post laminectomy pain, we have tried intraoperative perineural injection of lidocaine right after the exposure in expecting that this would be preemptive analgesia by blocking the nerve transmission so that postoperative pain starts later and lighter.

DETAILED DESCRIPTION:
A randomized double-blind 40 patients aged 18-50 of ASA I and II undergoing laminectomy were included in the study. All the patients were followed for their heart rate, arterial pressure , respiratory rate, oxygen saturation, end tidal CO2 and postoperative VAS scores.

All the patients were premedicated with midazolam 0.1 mg/kg intramuscularly 40 minutes prior to surgery. The induction was made 2 mg/kg propofol, 1 ug/kg remifentanyl, 0.5mg/kg rocuronium. After the orotracheal intubation anesthesia was maintained with isoflurane (%0.5-2.0) and 0.1 mg/kg rocuronium.Just before the exposure of dorsal root, 0.5 cc %2 lidocaine was injected on the dorsal root.The patients postoperative analgesic period, VAS scores and additional analgesic need was recorded. For the postoperative analgesia tramadol 1 mg/kg tramadol was used.

ELIGIBILITY:
Inclusion Criteria:

* laminectomy
* 18-50 age
* ASA 1-2
* both sex

Exclusion Criteria:

* under 18 or older than 50
* any disease other than back pain\
* ASA 3-4

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
In the laminectomy operation, right after the exposure of the dorsal root , an injection of lidocaine attenuates postoperative pain. | postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: cengiz Mordeniz, MD, Ass Prof, Study Chair — Harran University
Locations (1):
- harran University Education, Research and application hospital, Sanliurfa, Şanlıurfa, Turkey (Türkiye)